CLINICAL TRIAL: NCT04909931
Title: Vitamin D Supplementation on Outcome and Disease Activity in Rheumatoid Arthritis Patients At Rajavithi Hospital : a Randomized Clinical Trial
Brief Title: Vitamin D Supplementation on Outcome and Disease Activity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 64012
Record Dates: First submitted 2021-05-11; First posted 2021-06-02 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2022-02

CONDITIONS: Rheumatoid Arthritis, Vitamin D , Disease Activity, DAS28ESR
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Ergocalciferols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vitamin D supplementation group (Experimental): First arm ; add on vitamin D 40,000 IU/week for 12 weeks
  Interventions: Drug: Vitamin D 2
- second arm (Experimental): add on placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D 2 — Randomized allocation first arm : add on vitamin D supplementation 40,000 iu/week for 12 weeks
  Arms: vitamin D supplementation group
Drug: Placebo — Second arm : add on placebo for 12 weeks
  Arms: second arm

SUMMARY:
To study efficacy of Vitamin D on outcome and disease activity ; DAS28-ESR in Rheumatoid arthritis patients at Rajavithi hospital .

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yrs old
* RA diagnosed by ACR/EULAR 2010
* low to moderate disease activity
* on stable NSAIDs and DMARDs for at least 1 month
* Received Prednisolone less than or equal to 7.5 mg/day
* serum calcium, phosphorus and ALP are within normal limit.

Exclusion Criteria:

* Chronic kidney disease stage 3 or higher
* History of TB
* History of Chronic liver disease
* Pregnancy or breast-feeding
* adjustment of immuno-suppressive drugs, steroid
* other connective tissue disease
* Vitamin D allergy
* received other drugs which have vitamin D component
* serum Vitamin D less than 10 ng/mL

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
To study efficacy of vitamin D on disease activity RA patients at Rajavithi hospital | 12 weeks
  Determine disease activity by DAS28-ESR in relation with vitamin D supplementation.
To study efficacy of vitamin D on IL-6 in RA patients at Rajavithi hospital | 12 weeks
  DAS-28 ESR measure from swollen joint count, tender joint count, ESR and patient global assessment

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Nunthiyakul, Medicine, Study Chair — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Polasik K, Piotrowska E, Lipinska B, Witkowski JM, Bryl E, Tukaj S. Vitamin D status in patients with rheumatoid arthritis: a correlation analysis with disease activity and progression, as well as serum IL-6 levels. Acta Biochim Pol. 2017;64(4):667-670. doi: 10.18388/abp.2017_1636. Epub 2017 Dec 5. PMID 29202486
- [Background] Gopal K, Thevarajah M, Ng CM, Raja J. Effects of vitamin D on disease activity and serum interleukin-6 in rheumatoid arthritis. Int J Rheum Dis. 2019 May;22(5):834-841. doi: 10.1111/1756-185X.13484. Epub 2019 Feb 6. PMID 30729713
- [Background] Aslam MM, John P, Bhatti A, Jahangir S, Kamboh MI. Vitamin D as a Principal Factor in Mediating Rheumatoid Arthritis-Derived Immune Response. Biomed Res Int. 2019 May 7;2019:3494937. doi: 10.1155/2019/3494937. eCollection 2019. PMID 31205940